CLINICAL TRIAL: NCT04156464
Title: Phenobarbital Versus Ativan for Refractory Alcohol Withdrawal Treatment in the Intensive Care Unit
Brief Title: Phenobarbital vs Ativan for Alcohol Withdrawal in the Intensive Care Unit
Acronym: PARTI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Bhagat Aulakh, Principal Investigator, OSF Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1499413
Record Dates: First submitted 2019-10-16; First posted 2019-11-07 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Withdrawal; Alcohol Withdrawal Delirium
Keywords: lorazepam; phenobarbital; ativan; alcohol withdrawal syndrome; alcohol withdrawal; intensive care unit; delirium tremens; refractory alcohol withdrawal; benzodiazepine
MeSH Terms: conditions — Alcohol Withdrawal Delirium | interventions — Phenobarbital; Lorazepam

STUDY DESIGN:
Intervention Model Description: 2 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phenobarbital based treatment (Active Comparator): * The phenobarbital group will undergo management with a phenobarbital based treatment protocol with additional symptom triggered therapies.
  * On day 1, the phenobarbital group receive a loading dose of phenobarbital intravenous 10mg/kg (actual body weight) with a maximum dose of 1 g/100 mL
  * On day 2 of study protocol, and no sooner than 12 hours after loading dose, phenobarbital 64.8 mg is administered every 12 hours for two doses.
  * On day 3 of study protocol, patients will receive phenobarbital 32.4 mg every 12 hours for two doses.
  * On day 4 of study protocol, patients will receive phenobarbital 32.4 mg once, to be given 24 hours after last scheduled dose.
  * Throughout the 4 day protocol, the patient will have phenobarbital 65 mg every 6 hours as needed available either IM or IV, starting no sooner than 30 minutes after the loading dose.
  Interventions: Drug: Phenobarbital
- Lorazepam based treatment (Active Comparator): * The lorazepam group will undergo management with a lorazepam based treatment protocol with additional symptom triggered therapies.
  * On Day 1, the lorazepam group will be started on scheduled lorazepam 4 mg every 6 hours
  * After day 1, the scheduled lorazepam dose will be modified based on the total lorazepam requirements from the previous day and divided into 4-6 doses.
  * A lorazepam infusion, at physician discretion, will be available at any point if the dose of scheduled and PRN lorazepam being given is too high or frequent to effectively be administered.
  * Once symptoms are well controlled on lorazepam based therapy, the total dose given over the past 24 hours will be calculated and weaned by approximately 10-20% per day when clinically appropriate.
  * Throughout the entire protocol, 2-4 mg lorazepam IV q 30 minutes PRN will be available for a goal CIWA <6 or RASS -1 to 0.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Phenobarbital — Phenobarbital loading dose followed by a taper will be given to control acute alcohol withdrawal syndrome
  Other Names: solfoton; luminal
  Arms: Phenobarbital based treatment
Drug: Lorazepam — Ativan will be given according to our institutional alcohol withdrawal protocol to control acute alcohol withdrawal syndrome
  Other Names: ativan
  Arms: Lorazepam based treatment

SUMMARY:
Our aim is to compare outcomes of patients with benzodiazepine-refractory alcohol withdrawal syndrome who are treated with either a phenobarbital-based or a lorazepam based protocol.

DETAILED DESCRIPTION:
* This study is a prospective, open-label, randomized, controlled trial.
* The electronic medical record will be used to identify patients who have a diagnosis of alcohol withdrawal or are receiving alcohol withdrawal. Subjects who are anticipated to meet inclusion criteria will be pre-consented for the study using an informed consent process. see informed consent form.
* Subjects will not be enrolled and randomized until they have met inclusion criteria.
* If a patient meets criteria, but is deemed non-decisional or unable to give consent, the patient's medical decision maker will undergo the informed consent process.
* After enrollment, participants will be randomized to either the control group (lorazepam-based therapy) or the study group (phenobarbital-based therapy)
* Personnel unassociated with patient screening, enrollment, or follow up will create the allocation sequence and will use a random, computerized number generator. The allocation sequence will then be transferred to sequentially numbered, opaque envelopes for purposes of allocation concealment. These sequentially numbered envelopes, which are blinded to clinical trial coordinators/physicians, will be handed out in order as patients are enrolled. Clinical trial coordinators/physicians will verify treatment eligibility and informed consent before opening the envelope to obtain the treatment assignment.
* The study group will be placed on the phenobarbital-based protocol as described below in procedures. The control group will be placed on the lorazepam-based protocol, also listed below in procedures.
* All medications in the study are FDA approved. No investigational medicines will be used.
* Data will be collected on each participant as noted below in measurements.
* The data will be analyzed and published as noted above in the statistical analysis plan and data use and management section.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for randomization if he/she has met one of the following three conditions:

  1. has required more than 10 mg of lorazepam within a one hour time period,
  2. has required more than 30 mg of lorazepam within a four hour time period, or
  3. requires admission/transfer to the intensive care unit for primarily uncontrolled alcohol withdrawal symptoms

     Exclusion Criteria:
* Patients will be excluded from the study if he/she:

  1. has a traumatic brain injury or other neurological condition requiring frequent neurological assessment (stroke, intracranial hemorrhage, active seizures on admission)
  2. has severe hypotension requiring vasopressor support
  3. is less than 18 years of age
  4. is actively pregnant
  5. has an allergy to either of the drugs being studied (phenobarbital or lorazepam)
  6. is already intubated at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
ICU length of stay | study completion, up to 18 months
  number of days in the intensive care unit

SECONDARY OUTCOMES:
Hospital length of stay | Study completion, up to 18 months
  number of days in the hospital
30-day readmission | study complettion, up to 18 months
  rate of readmission of patients within 30 days for any cause
mortality | Study completion, up to 18 months
  number of deaths
Intubation | study completion, up to 18 months
  rate of endotracheal intubation
Hospitalization cost | Study completion, up to 18 months
  Cost of index hospital stay
Lorazepam use | Study completion, up to 18 months
  total lorazepam use in mg during the entire hospital stay
dexmedetomidine use | Study completion, up to 18 months
  total dexmedetomidine used in mcg during the entire hospital stay
propofol use | Study completion, up to 18 months
  total propofol used in mg during the entire hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Bhagat Aulakh, MD, Principal Investigator — OSF Healthcare System
Locations (1):
- OSF Saint Francis Medical Center, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedmann PD. Alcohol use in adults. N Engl J Med. 2013 Apr 25;368(17):1655-6. doi: 10.1056/NEJMc1302445. No abstract available. PMID 23614598
- [Background] Saitz R, Friedman LS, Mayo-Smith MF. Alcohol withdrawal: a nationwide survey of inpatient treatment practices. J Gen Intern Med. 1995 Sep;10(9):479-87. doi: 10.1007/BF02602395. PMID 8523149
- [Background] Kosten TR, O'Connor PG. Management of drug and alcohol withdrawal. N Engl J Med. 2003 May 1;348(18):1786-95. doi: 10.1056/NEJMra020617. No abstract available. PMID 12724485
- [Background] Holbrook AM, Crowther R, Lotter A, Cheng C, King D. Diagnosis and management of acute alcohol withdrawal. CMAJ. 1999 Mar 9;160(5):675-80. PMID 10102003
- [Background] Miller NS, Gold MS. Management of withdrawal syndromes and relapse prevention in drug and alcohol dependence. Am Fam Physician. 1998 Jul;58(1):139-46. PMID 9672434
- [Background] Kaim SC, Klett CJ, Rothfeld B. Treatment of the acute alcohol withdrawal state: a comparison of four drugs. Am J Psychiatry. 1969 Jun;125(12):1640-6. doi: 10.1176/ajp.125.12.1640. No abstract available. PMID 4890289
- [Background] Sarff M, Gold JA. Alcohol withdrawal syndromes in the intensive care unit. Crit Care Med. 2010 Sep;38(9 Suppl):S494-501. doi: 10.1097/CCM.0b013e3181ec5412. PMID 20724883
- [Background] Dixit D, Endicott J, Burry L, Ramos L, Yeung SY, Devabhakthuni S, Chan C, Tobia A, Bulloch MN. Management of Acute Alcohol Withdrawal Syndrome in Critically Ill Patients. Pharmacotherapy. 2016 Jul;36(7):797-822. doi: 10.1002/phar.1770. Epub 2016 Jun 30. PMID 27196747
- [Background] Hack JB, Hoffmann RS, Nelson LS. Resistant alcohol withdrawal: does an unexpectedly large sedative requirement identify these patients early? J Med Toxicol. 2006 Jun;2(2):55-60. doi: 10.1007/BF03161171. PMID 18072114
- [Background] Wong A, Benedict NJ, Lohr BR, Pizon AF, Kane-Gill SL. Management of benzodiazepine-resistant alcohol withdrawal across a healthcare system: Benzodiazepine dose-escalation with or without propofol. Drug Alcohol Depend. 2015 Sep 1;154:296-9. doi: 10.1016/j.drugalcdep.2015.07.005. Epub 2015 Jul 16. PMID 26205315
- [Background] Duby JJ, Berry AJ, Ghayyem P, Wilson MD, Cocanour CS. Alcohol withdrawal syndrome in critically ill patients: protocolized versus nonprotocolized management. J Trauma Acute Care Surg. 2014 Dec;77(6):938-43. doi: 10.1097/TA.0000000000000352. PMID 25248063
- [Background] Crispo AL, Daley MJ, Pepin JL, Harford PH, Brown CV. Comparison of clinical outcomes in nonintubated patients with severe alcohol withdrawal syndrome treated with continuous-infusion sedatives: dexmedetomidine versus benzodiazepines. Pharmacotherapy. 2014 Sep;34(9):910-7. doi: 10.1002/phar.1448. Epub 2014 Jun 5. PMID 24898418
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Ives TJ, Mooney AJ 3rd, Gwyther RE. Pharmacokinetic dosing of phenobarbital in the treatment of alcohol withdrawal syndrome. South Med J. 1991 Jan;84(1):18-21. doi: 10.1097/00007611-199101000-00006. PMID 1986421
- [Background] Tangmose K, Nielsen MK, Allerup P, Ulrichsen J. Linear correlation between phenobarbital dose and concentration in alcohol withdrawal patients. Dan Med Bull. 2010 Aug;57(8):A4141. PMID 20682131
- [Background] Kramp P, Rafaelsen OJ. Delirium tremens: a double-blind comparison of diazepam and barbital treatment. Acta Psychiatr Scand. 1978 Aug;58(2):174-90. doi: 10.1111/j.1600-0447.1978.tb06930.x. PMID 358756
- [Background] Martin PR, Bhushan CM, Kapur BM, Whiteside EA, Sellers EM. Intravenous phenobarbital therapy in barbiturate and other hypnosedative withdrawal reactions: a kinetic approach. Clin Pharmacol Ther. 1979 Aug;26(2):256-64. doi: 10.1002/cpt1979262256. PMID 455894
- [Background] Robinson GM, Sellers EM, Janecek E. Barbiturate and hypnosedative withdrawal by a multiple oral phenobarbital loading dose technique. Clin Pharmacol Ther. 1981 Jul;30(1):71-6. doi: 10.1038/clpt.1981.129. PMID 7237901
- [Background] Young GP, Rores C, Murphy C, Dailey RH. Intravenous phenobarbital for alcohol withdrawal and convulsions. Ann Emerg Med. 1987 Aug;16(8):847-50. doi: 10.1016/s0196-0644(87)80520-6. PMID 3619162
- [Background] Hendey GW, Dery RA, Barnes RL, Snowden B, Mentler P. A prospective, randomized, trial of phenobarbital versus benzodiazepines for acute alcohol withdrawal. Am J Emerg Med. 2011 May;29(4):382-5. doi: 10.1016/j.ajem.2009.10.010. Epub 2010 Mar 25. PMID 20825805
- [Background] Rosenson J, Clements C, Simon B, Vieaux J, Graffman S, Vahidnia F, Cisse B, Lam J, Alter H. Phenobarbital for acute alcohol withdrawal: a prospective randomized double-blind placebo-controlled study. J Emerg Med. 2013 Mar;44(3):592-598.e2. doi: 10.1016/j.jemermed.2012.07.056. Epub 2012 Sep 19. PMID 22999778
- [Background] Ibarra F Jr. Single dose phenobarbital in addition to symptom-triggered lorazepam in alcohol withdrawal. Am J Emerg Med. 2020 Feb;38(2):178-181. doi: 10.1016/j.ajem.2019.01.053. Epub 2019 Jan 30. PMID 30744913
- [Background] Tidwell WP, Thomas TL, Pouliot JD, Canonico AE, Webber AJ. Treatment of Alcohol Withdrawal Syndrome: Phenobarbital vs CIWA-Ar Protocol. Am J Crit Care. 2018 Nov;27(6):454-460. doi: 10.4037/ajcc2018745. PMID 30385536
- [Background] Gold JA, Rimal B, Nolan A, Nelson LS. A strategy of escalating doses of benzodiazepines and phenobarbital administration reduces the need for mechanical ventilation in delirium tremens. Crit Care Med. 2007 Mar;35(3):724-30. doi: 10.1097/01.CCM.0000256841.28351.80. PMID 17255852
- [Background] Gashlin LZ, Groth CM, Wiegand TJ, et al. Comparison of alcohol withdrawal outcomes in patients treated with benzodiazepines alone versus adjunctive phenobarbital: a retrospective cohort study. Asia Pac J Med Toxicol 2015;4:31-6.
- [Background] Hjermo I, Anderson JE, Fink-Jensen A, Allerup P, Ulrichsen J. Phenobarbital versus diazepam for delirium tremens--a retrospective study. Dan Med Bull. 2010 Aug;57(8):A4169. PMID 20682133
- [Background] Askgaard G, Hallas J, Fink-Jensen A, Molander AC, Madsen KG, Pottegard A. Phenobarbital compared to benzodiazepines in alcohol withdrawal treatment: A register-based cohort study of subsequent benzodiazepine use, alcohol recidivism and mortality. Drug Alcohol Depend. 2016 Apr 1;161:258-64. doi: 10.1016/j.drugalcdep.2016.02.016. Epub 2016 Feb 18. PMID 26922279
- [Background] Mo Y, Thomas MC, Karras GE Jr. Barbiturates for the treatment of alcohol withdrawal syndrome: A systematic review of clinical trials. J Crit Care. 2016 Apr;32:101-7. doi: 10.1016/j.jcrc.2015.11.022. Epub 2015 Dec 8. PMID 26795441